CLINICAL TRIAL: NCT03777527
Title: My PICU Diary: a Patient Diary for Critically Ill Children
Brief Title: PICU Patient Diary
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Other Study IDs: 5843
Record Dates: First submitted 2018-12-13; First posted 2018-12-17 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The PICU-Diary study is a prospective single centre pilot study in the Pediatric Critical Care Unit at McMaster Children's Hospital. We will evaluate the impressions of family caregivers and healthcare providers on the PICU Patient Diary, and its acceptability for use in the PICU, using mixed methods. We will assess the feasibility of assessing the impact of a patient diary on PICU outcomes and psychological distress in critically ill children, 1 month following PICU discharge.

DETAILED DESCRIPTION:
There is considerable need for research dedicated to exploring interventions to improve the psychological and functional effects of critical care admission on patients and families. Patient diaries are one approach that has been used in several adult critical care groups and has been shown to positively impact patient care by helping patients better understand their illness, acting as a therapeutic tool and debriefing aid, and providing an outlet for caregivers to participate in care plans. However, to date, there is minimal research available in the pediatric population.

The specific objectives of this study are to evaluate the acceptability and impressions of a patient diary as a supportive measure for critically ill children in the PICU. Our secondary objective is to evaluate the feasibility of measuring the impact of a patient diary on psychological distress in critically ill children, following discharge from the PICU.

The purpose of this diary is to support the recovery of critically ill children and their family members by:

1. Helping patients understand visually and in written form as age appropriate, what has happened to them during their PICU stay, how ill they were, and in so doing, reduce anxiety and post-traumatic stress symptoms; AND
2. Serving as an engagement tool to help families take on an informed, active role in their child's care plan.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients admitted to the PICU will be screened for eligibility to participate in the evaluation component of the PICU Diary study
* We will offer a PICU Diary to families of any critically ill children admitted to the PICU for at least 72 hours and who are fluent in the English language
* Eligible patients and their families will be approached for consent to participate, by a member of the investigator team (MB, KC, SB or CC). For those who consent to participate, they will be oriented to the diary and its use.

Exclusion Criteria:

* Stay less than 72 hours
* Not fluent in the English language

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Critically ill patients and their families admitted to the PICU at McMaster Children's Hospital
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Patient Diary Acceptability | 1 day
  Acceptability of the diary to family members, patients, and healthcare providers in the PICU to determine the perception of impact of the diary on patient recovery. Information collected with surveys and qualitative interviews.
Feasability of measuring psychological well-being | 1 day
  Patient reported outcome measure of psychological well-being after critical illness with Children's Critical Illness Impact Scale

CONTACTS AND LOCATIONS:
Overall Officials: Karen Choong, MD, Principal Investigator — McMaster University
Locations (1):
- McMaster Children's Hospital, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No